CLINICAL TRIAL: NCT01427543
Title: The HJ MILE HIV Prevention Intervention for Post-incarcerated Bisexual African American Men
Brief Title: The HJ MILE HIV Prevention Intervention for Post-incarcerated Men
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Charles Drew University of Medicine and Science (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ricky Bluthenthal, Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HS-10-00590; 5UR6PS001098 (NIH)
Record Dates: First submitted 2011-08-30; First posted 2011-09-01 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: HIV; Risk Reduction Behavior
Keywords: behavioral intervention; HIV risk reduction; African Americans; incarceration; bisexual; reduce risk behaviors
MeSH Terms: conditions — Risk Reduction Behavior; Bisexuality

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MILE group sessions (Experimental): Participants will attend 6 - 2 hour long, interactive, culturally congruent, group sessions that address knowledge, beliefs, attitudes, and skills related to reducing HIV risk behaviors.
  Interventions: Behavioral: MILE intervention
- Control (No Intervention): These subjects will be provided with access to post-incarcerations services that will be provided by the Center for Health Justice.

INTERVENTIONS:
Behavioral: MILE intervention — Participants will be asked to attend 6 - 2 hour group sessions over the course of 3 weeks. The intervention aims to reduce HIV risk taking related to sex risk and alcohol and drug use.
  Arms: MILE group sessions

SUMMARY:
The goal of this study is to determine whether a culturally congruent, group intervention can reduce HIV risk behaviors among recently incarcerated, bisexual, African American men.

DETAILED DESCRIPTION:
The goal of this study is to evaluate the efficacy of the Men in Life Environments (MILE) intervention, adapted from the Men of African American Legacy Empowering Self (MAALES) Project, an innovative and culturally congruent intervention designed to reduce HIV risk-related behaviors and improve psychosocial outcomes in recently incarcerated African American men who have sex with men and women (MSMW). The MILE intervention is guided by the Theory of Reasoned Action and Planned Behavior, the Critical Thinking and Cultural Affirmation (CTCA) Model, and the Empowerment Theory. The small group MILE intervention involves six two-hour group sessions held over three weeks and is lead by two African-American co-facilitators. The investigators will test the intervention with a total of 260 African American MSMW, evenly randomized to intervention and control conditions. For this study, participants will be interviewed at baseline, shortly after completion of the intervention (~ 4 weeks after baseline), and again 3 months following the second interview. This project will be among the first to develop and test an HIV risk-reduction intervention designed specifically for African American post-incarcerated MSMW. Study aims are as follows:

Aim 1: To evaluate the impact of the MILE intervention on rates of condom use, having sex while under the influence of drugs and alcohol, and number of sex partners among recently incarcerated bisexual African American MSMW.

Hypothesis: Compared to the control condition, the MILE intervention condition will be more effective in decreasing episodes of unprotected anal and vaginal intercourse, incidents of sex under the influence of drugs and alcohol and numbers of intercourse partners at the 3-month follow-up assessment.

Aim 2: To evaluate the impact of the MILE intervention on uptake of testing for sexually transmitted infections (STI) among recently incarcerated African American MSMW.

Hypothesis: Compared to the control condition, the MILE intervention participants will be more likely to accept STI testing after the post-intervention assessment.

Aim 3: To describe social support and social networks of recently incarcerated African American MSMW and to examine whether these factors are associated with HIV risk in this population.

The MILE intervention will be implemented by The Center for Health Justice (CHJ) - a community-based HIV prevention and care advocacy organization that has been working with incarcerated and post-incarcerated populations since 1997. The adaptation and implementation of this intervention by CHJ should increase the dissemination and applicability of the intervention to other locales should it prove to be effective.

ELIGIBILITY:
Inclusion Criteria:

* self-identified as African American or Black
* male
* 18 years of age or greater
* Los Angeles County resident
* Been incarcerated in the last 12 months
* oral or anal sex with a man in the last 12 months
* any unprotected anal or vaginal sex in the last 3 months
* two or more sex partners in the last 3 months

Exclusion Criteria:

* Female or transgendered
* not self-identified as African American or Black
* any self-reported illicit drug injection in the last 12 months

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2011-07; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Condom use | Last 3 months
  This measure captures the percentage of times that participants self-report using a condom during vaginal and anal sex.
Sex under the influence of alcohol and drugs | Last 3 months
  Self-reported vaginal or anal sex while under the influence of alcohol or drugs.
Number of sex partners | Last 3 month
  Participant's self-report of number of sex partners in the last 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Ricky Bluthenthal, Ph.D., Principal Investigator — University of Southern California
Locations (1):
- Center for Health Justice, Los Angeles, California, United States

REFERENCES:
- [Result] Dangerfield DT 2nd, Harawa NT, Smith LR, Jeffries WL 4th, Baezconde-Garbanati L, Bluthenthal R. Latent Classes of Sexual Risk Among Black Men Who Have Sex with Men and Women. Arch Sex Behav. 2018 Oct;47(7):2071-2080. doi: 10.1007/s10508-017-1142-y. Epub 2018 Mar 14. PMID 29541914
- [Result] Harawa NT, Guentzel-Frank H, McCuller WJ, Williams JK, Millet G, Belcher L, Joseph HA, Bluthenthal RN. Efficacy of a Small-Group Intervention for Post-Incarcerated Black Men Who Have Sex with Men and Women (MSMW). J Urban Health. 2018 Apr;95(2):159-170. doi: 10.1007/s11524-018-0227-9. PMID 29541962
- [Result] Joseph HA, Pan Y, Mendoza M, Harawa NT, Lauby J, Hosek SG, Bluthenthal RN, Milnamow M, Fernandez MI, Jeffries WL 4th, Belcher L, Millett GA. HIV Acquisition and Transmission Potential Among African American Men Who Have Sex with Men and Women in Three U.S. Cities. Arch Sex Behav. 2018 Jan;47(1):183-194. doi: 10.1007/s10508-017-1052-z. Epub 2017 Nov 9. PMID 29124541
- [Result] Li MJ, Frank HG, Harawa NT, Williams JK, Chou CP, Bluthenthal RN. Racial Pride and Condom Use in Post-Incarcerated African-American Men Who Have Sex With Men and Women: Test of a Conceptual Model for the Men in Life Environments Intervention. Arch Sex Behav. 2018 Jan;47(1):169-181. doi: 10.1007/s10508-016-0734-2. Epub 2016 Apr 26. PMID 27115618